CLINICAL TRIAL: NCT01096017
Title: A Study to Investigate the Relative Efficacy of Terbutaline Turbuhaler® 0.4 mg and Salbutamol Pressurized Metered Dose Inhaler (pMDI) 200 μg - a Single Blind, Single Dose, Randomized, Crossover, Phase III Study in Japanese Adult Asthma Patients
Brief Title: To Investigate the Relative Efficacy of Terbutaline Turbuhaler® and Salbutamol Pressurized Metered Dose Inhaler (pMDI) a Single Blind Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D589LC00002
Record Dates: First submitted 2010-03-19; First posted 2010-03-30 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Terbutaline; Turbuhaler; Efficacy; Asthma; Japanese; salbutamol; Bricanyl
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Terbutaline Turbuhaler® 0.4mg + pMDI placebo pMDI ⇒salbutamol pMDI 200 μg +placebo Turbuhaler®
  Interventions: Drug: Terbutaline Turbuhaler®; Other: pMDI placebo pMDI; Other: Placebo Turbuhaler®
- 2 (Experimental): salbutamol pMDI 200 μg +placebo Turbuhaler® ⇒Terbutaline Turbuhaler® 0.4mg + pMDI placebo pMDI
  Interventions: Drug: Salbutamol pMDI; Other: pMDI placebo pMDI; Other: Placebo Turbuhaler®

INTERVENTIONS:
Drug: Terbutaline Turbuhaler® — 0.4 mg, inhalation, single dose
  Other Names: Bricanyl Turbuhaler
  Arms: 1
Drug: Salbutamol pMDI — 200 μg, inhalation, single dose
  Other Names: Saltanol
  Arms: 2
Other: pMDI placebo pMDI — Placebo pMDI 2 inhalations
Other: Placebo Turbuhaler® — Placebo Turbuhaler 1 inhalation

SUMMARY:
This is a single blind, single dose, crossover study to investigate the relative efficacy of terbutaline Turbuhaler® 0.4 mg in relation to salbutamol pressurized Metered Dose Inhaler (pMDI) 200 μg in Japanese adult asthmatic patients.The secondary objective of this study is to investigate safety of terbutaline Turbuhaler® 0.4 mg in Japanese adult asthma patients by means of adverse events (AEs) and vital signs (blood pressure, pulse rate). The subject population includes Japanese patients (16 years of age or older) with asthma who need treatment with inhaled Glucocorticosteroids (ICS).

ELIGIBILITY:
Inclusion Criteria:

* On ICS for at least 3 months from Visit 2 and with a prescribed constant dose during the 4 weeks prior to Visit 2
* Forced Expiratory Volume in 1 Second (FEV1) of at least 50 % of predicted normal value pre-bronchodilator
* Reversible airway obstruction according to reversibility test performed at Visit 2, defined as an increase in Forced Expiratory Volume in 1 Second (FEV1) ≥12% relative baseline at 15-30 minutes after inhalation of in total 400 μg salbutamol

Exclusion Criteria:

* Treatment with oral, parenteral or rectal GCS (Glucocorticosteroids)within 4 weeks or depot parenteral GCS (Glucocorticosteroids) within 3 months prior to Visit 2.
* Change in prescribed asthma medication due to exacerbation of asthma within 4 weeks prior to Visit 2 or being hospitalized due to exacerbation of asthma within 8 weeks prior to Visit 2.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Chair — AstraZeneca
Locations (1):
- Research Site, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited at one clinic in Tokyo, Japan, between March and April 2010
Pre-assignment Details: 37 participants enrolled; 13 excluded (9 due to eligibility criteria not fulfilled and 4 for other reasons)
Groups:
- Salbutamol First, Then Terbutaline: Salbutamol pMDI 200 μg +placebo Turbuhaler® ⇒Terbutaline Turbuhaler® 0.4mg + pMDI placebo pMDI
- Terbutaline First, Then Salbutamol: Terbutaline Turbuhaler® 0.4mg + pMDI placebo pMDI ⇒Salbutamol pMDI 200 μg +placebo Turbuhaler®
Period: Treatment Period 1
Arm/Group | Salbutamol First, Then Terbutaline | Terbutaline First, Then Salbutamol
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout 1 - 14 Days
Arm/Group | Salbutamol First, Then Terbutaline | Terbutaline First, Then Salbutamol
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Salbutamol First, Then Terbutaline | Terbutaline First, Then Salbutamol
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Eligibility criteria not fulfilled | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) Area Under Curve (AUC) 0-4 Hours After Drug Inhalation
Description: FEV1 (Forced Expiratory Volume in 1 second) AUC 0-4 hours after drug inhalation
Time Frame: At two visits during a maximum of 15 days. FEV1 timepoints: all time points t=5, 15, 30, 60, 120, 180 and 240 minutes.
Measure: Geometric Mean (Full Range); unit: milliLiters x minutes
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
milliLiters x minutes | 617.56 [352.57 to 974.45] | 634.64 [356.68 to 1016.46]

2. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 5 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 115.58 [102.80 to 137.95] | 112.80 [100.00 to 134.85]

3. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 15 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 118.15 [105.11 to 142.16] | 115.69 [103.27 to 138.59]

4. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 30 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 119.42 [103.28 to 147.32] | 117.02 [99.59 to 139.83]

5. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 60 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 120.28 [102.19 to 149.19] | 118.11 [102.86 to 144.40]

6. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 120 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 119.54 [97.45 to 149.73] | 119.79 [103.27 to 150.21]

7. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 180 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 116.68 [92.70 to 142.70] | 118.48 [100.68 to 146.06]

8. Secondary Outcome: FEV1 (Forced Expiratory Volume in 1 Second) at 240 Minutes After Inhalations of Study Drug as Percentage of Pre-dose
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percentage of Pre-Dose FEV1
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percentage of Pre-Dose FEV1 | 113.59 [87.96 to 132.67] | 117.05 [97.96 to 139.00]

9. Secondary Outcome: Maximum % Change in FEV1 (Forced Expiratory Volume in 1 Second) Within 4 Hours After Drug Inhalation
Description: percent of pre-dose (ratio)
Time Frame: At two visits during a maximum of 15 days
Measure: Geometric Mean (Full Range); unit: Percent change
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Percent change | 122.62 [105.11 to 149.73] | 121.43 [105.31 to 150.21]

10. Secondary Outcome: Time to Peak FEV1 (Forced Expiratory Volume in 1 Second) Within 4 Hours After Drug Inhalation
Description: Time to peak measurement of FEV1 (min)
Time Frame: At two visits during a maximum of 15 days
Measure: Median (Full Range); unit: Minutes
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Minutes | 60.00 [5.00 to 180.00] | 120.00 [5.00 to 240.00]

11. Secondary Outcome: Number of Patients With % Change in FEV1 (Forced Expiratory Volume in 1 Second) >15% Within 4 Hours After Drug Inhalation
Description: Number of patients with % change in FEV1 >15% within 4 hours after drug inhalation.
Time Frame: At two visits during a maximum of 15 days
Measure: Number; unit: Participants
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Participants | 17 | 16

12. Secondary Outcome: Time to Change More Than or Equal to 15% (Time to Onset Response) Within 4 Hours After Drug Inhalation
Description: Time to change more than or equal to 15% (time to onset response) within 4 hours after drug inhalation
Time Frame: At two visits during a maximum of 15 days
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Number analyzed (Participants) | 22 | 22
Minutes | 31.36 (37.49) | 34.32 (40.31)

ADVERSE EVENTS:
Arm/Group | Salbutamol pMDI | Terbutaline Turbuhaler®
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less